CLINICAL TRIAL: NCT07173465
Title: Comparison of the Effects of Physical Activity and Virtual Reality Training on Physical Function, Cognition and Quality of Life in Patients With Schizophrenia
Brief Title: Comparison of the Effects of Physical Activity and Virtual Reality Training in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 64-2023
Record Dates: First submitted 2023-05-25; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Balance; Distorted; Cognitive Impairment
Keywords: schizophrenia; Virtual reality; Cognition
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Exercise; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Activity (PA group) (Active Comparator): The program will be comprised of
  (5 minutes) Warm-up (5 minutes) Strengthening exercises (Lunges- squats) (10 minutes) Balance and Cardiovascular endurance (HIIT-penguin seesaw- table tilt) (15 minutes) Aerobic ex (stationary bike- dancing) (5 minutes) Cool down exercises and breathing control. In addition to all these, the individuals will continue occupational therapy.
  Interventions: Device: Virtual Reality (VR)
- Virtual Reality (VR) group (Active Comparator): Group 2 Virtual Reality (VR) group will undergo 45 minutes of the Nintendo Wii-FitTM game. First of all, it will start with games that include warm-up exercises ( 5 min) and then continue with games that include strengthening (5 min), balance (5 min) and aerobic exercises (15 min).
  Finally, the treatment will be terminated with games, including cool-down (5 min) exercises. In addition to all these, the individuals will continue occupational therapy.
  Interventions: Other: Physical Activity (PA group)
- control group (Sham Comparator): This group will undergo regular occupational therapy at the treatment center
  Interventions: Other: occupational therapy

INTERVENTIONS:
Device: Virtual Reality (VR) — Participants will engage in the VR gaming intervention three times a week for 12 weeks. Each session will last approximately 45 minutes, providing ample gameplay, instruction, and debriefing time.
  Arms: Physical Activity (PA group)
Other: Physical Activity (PA group) — The intervention includes a 5-minute warm-up, 10 minutes of strengthening exercises (lunges and squats), 20 minutes of balance and cardiovascular endurance activities (HIIT exercises), 20 minutes of aerobic exercises (stationary bike and dancing), and a 5-minute cool-down with breathing control. Participants also continue with personalized occupational therapy to enhance their functional abilities.
  Arms: Virtual Reality (VR) group
Other: occupational therapy — the group will undergo their normal occupational therapy activities that include drawing, coloring, mathematical problems as well as solving mazes
  Arms: control group

SUMMARY:
The current study aims to compare the effects of physical activity and Virtual Reality training on physical function, cognition and quality of life in patients with Schizophrenia.

It is hypothesized in the literature that both physical activity and VR may have positive effects on the symptoms of PwS. Still, which modality may be more effective has yet to be discovered. By comparing the effects of physical activity and VR training on the symptoms of PwS, this study may provide valuable insights into the potential benefits of these interventions and inform the development of effective treatment strategies for PwS.

Our study will discuss this relationship, and the results will be presented.

DETAILED DESCRIPTION:
1 INTRODUCTION AND PURPOSE

Schizophrenia is a debilitating mental disorder characterized by disruptions in thinking, perception, emotions, and social functioning (1). Patients with schizophrenia (PwS) often experience impairments in physical function, cognition, and quality of life, which can significantly impact their overall well-being. As part of the pursuit to enhance treatment outcomes, researchers, including physical therapists, have explored various adjunctive therapies that can potentially alleviate these impairments. In this study, we aim to compare the effects of physical activity (PA) and virtual reality (VR) training on physical function, cognition, and quality of life in Patients with schizophrenia (PwS), compared to a control group that undergoes regular occupational therapy.

1.1 Background Physical activity has been recognized as a beneficial intervention for individuals with mental disorders, including schizophrenia (2). Engaging in regular physical activity has been associated with improved physical fitness, cardiovascular health, and muscle strength. Furthermore, studies have shown that physical activity can positively influence cognitive function, including attention, memory, and executive functions, in individuals with schizophrenia (2, 3). These improvements in physical and cognitive domains can potentially lead to enhanced quality of life for these individuals.

Virtual reality training, on the other hand, is an emerging therapeutic approach that provides immersive and interactive experiences through computer-generated simulations. While the benefits of physical activity have been extensively studied in schizophrenia, research investigating the specific effects of virtual reality training in this population is limited (4). There is a need to explore the potential benefits of VR in improving physical function, cognition, and quality of life in individuals with schizophrenia to expand our understanding of its therapeutic value.

1.2 Significance Understanding the comparative effects of physical activity and virtual reality training on physical function, cognition, and quality of life in Patients with schizophrenia (PwS), in comparison to the control group undergoing regular occupational therapy, holds significant importance. By comparing these interventions, we can identify their relative effectiveness and potential benefits in addressing the impairments associated with schizophrenia. This knowledge can inform clinicians, researchers, and healthcare professionals, including physical therapists, in making evidence-based decisions regarding the use of these interventions in clinical practice. Additionally, it may contribute to the development of personalized treatment approaches that optimize outcomes and improve the overall well-being of individuals with schizophrenia.

1.3 Overview This study describes a comparative analysis of three groups: a physical activity intervention group, a virtual reality training intervention group, and a control group that undergoes regular occupational therapy at the center. The study will recruit a sample of individuals diagnosed with schizophrenia and randomly assign them to one of the three groups. Assessments of physical function, cognitive performance, and quality of life will be conducted before and after the interventions to evaluate the effectiveness of each approach. The findings of this study will contribute to the existing literature and inform the development of evidence-based interventions for individuals with schizophrenia, particularly in the context of physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20 and 77 years old.
* Willing to participate in research.
* Diagnosed with Schizophrenia according to the criteria defined in the DSM-IV by a psychiatrist.
* Able to attend Community Mental Health Center regularly.
* Not diagnosed with a mental disability, alcoholism, or drug addiction.
* Scoring 40 points or higher on the GAF test, indicating a non-severe mental state.
* Capable of fully understanding the purpose and content of the research.
* Able to participate in physical activity that requires musculoskeletal movement without difficulty, as determined by self-report.

Exclusion Criteria:

* Have significant cardiovascular, neuromuscular, endocrine, or other disorders that might prevent safe participation in the study.
* Have a diagnosis of alcohol or substance abuse.
* Have a secondary diagnosis of neurological disease or disease associated with the consumption of toxins, addiction to technology, or compulsive gambling.
* Unable to read, understand, or respond to assessment tests.

Ages: 20 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Simple Physical Activity Questionnaire | 12 weeks
  The SIMPAQ is a five-point evaluation tool designed to assess physical activity and sedentary behavior in individuals with common mental disorders.
Six minute walking test | 12 weeks
  The 6-Minute Walk Test (6MWT) is a standardized physical performance test that measures the distance an individual can walk on a flat, hard surface in six minutes. It provides an objective assessment of functional exercise capacity, endurance, and overall mobility in daily life activities.
The Mini-Mental State Examination | 12 weeks
  The Mini-Mental State Examination (MMSE) is commonly used as a screening tool to assess cognitive function and detect cognitive impairments. While the MMSE is not specifically designed to evaluate cognitive deficits associated with schizophrenia, it can still provide some insights into general cognitive functioning in individuals with schizophrenia.
  In schizophrenia, cognitive impairments are frequently observed across various cognitive domains, including attention, working memory, executive function, verbal fluency, and processing speed. These cognitive deficits can significantly impact daily functioning, quality of life, and overall outcomes for individuals with schizophrenia.
SF-36 | 12 weeks
  It is a widely used self-report questionnaire that assesses health-related quality of life (HRQoL)
Berg Balance Scale | 12 weeks
  Berg Balance Scale (BBS) is a standardized clinical test used to evaluate static and dynamic balance. It consists of 14 functional tasks, such as standing, reaching, and turning, each scored on a 5-point scale. The total score provides an objective measure of balance performance and fall risk in individuals.
Time Up and Go Test | 12 weeks
  The Timed Up and Go Test (TUG) is a standardized assessment that measures functional mobility. Participants are asked to stand up from a seated position, walk three meters, turn around, walk back, and sit down. The time taken to complete the task is recorded, providing an objective measure of mobility, balance, walking ability, and fall risk
Sit to Stand test | 12 weeks
  "The Sit-to-Stand Test is a functional performance measure used to assess lower limb strength, endurance, and mobility. Participants are asked to rise from a seated position to a full stand and return to sitting, repeated either for a set number of repetitions (e.g., five times) or within a fixed time period (e.g., 30 seconds). The total time or number of repetitions provides an objective indicator of lower body function and fall risk.
Grip strength | 12 weeks
  he Grip Strength Test is a standardized assessment of hand and forearm muscle strength. Participants are instructed to squeeze a calibrated hand dynamometer with maximum effort, usually in a seated position with the elbow at 90 degrees. The highest value from repeated trials is recorded, providing an objective measure of upper extremity strength and overall functional capacity

SECONDARY OUTCOMES:
Calgary Depression Scale | 12 weeks
  The Calgary Depression Scale was developed by Addington et al. (1994) as a tool to measure the presence and severity of depressive symptoms in patients with schizophrenia.
Katz Activities of Daily Living Scale | 12 weeks
  The Katz Index of Independence in ADLs (Katz Index) is a widely used tool to assess basic activities of daily living (ADLs) such as bathing, dressing, toileting, transferring, continence, and feeding.
Lawton Brody Instrumental Activities of Daily Living Scale | 12 weeks
  IADL is a commonly used tool to assess the level of independence in instrumental activities of daily living in older adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No